CLINICAL TRIAL: NCT03410667
Title: A Patient-centered Approach to Urinary Incontinence and Quality of Life in Children and Adolescents With Spina Bifida
Brief Title: Incontinence and Quality of Life in Children With Spina Bifida
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Konrad Szymanski, Assistant Professor of Urology, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1707207063; 5K23DK119368 (NIH)
Record Dates: First submitted 2017-12-13; First posted 2018-01-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Spina Bifida; Myelomeningocele
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Other): Standard of care arm
  Interventions: Behavioral: Phase One: Exploration; Behavioral: Phase Two: Creation; Behavioral: Phase Three: Reflection
- Intervention Arm (Experimental): Intervention arm
  Interventions: Behavioral: Aim 3

INTERVENTIONS:
Behavioral: Phase One: Exploration — Spina Bifida patients from the pediatric urology clinic at Riley Hospital and their caregivers will participate in discussions of UI goals. These patients will self report their experiences and perspectives using a "Day in the Life" diary tool-kit.
  Arms: Standard Care
Behavioral: Phase Two: Creation — Patients, caregivers and providers will work to create a goal setting tool to help patients and physicians appropriately address the issue of UI in patients with spina bifida.
  Arms: Standard Care
Behavioral: Phase Three: Reflection — This is a validation step to test whether the goal-setting tool is widely applicable and functional in a clinic setting. There will be cognitive interviews after the tool is completed to gather patient impressions.
  Arms: Standard Care
Behavioral: Aim 3 — This will be a large scale validation of the app, with assignment to standard care for the first year of enrollment.
  Other Names: Prospective Assessment of Patient-Centered Goals and HRQOL
  Arms: Intervention Arm

SUMMARY:
This study aims to develop an innovative, interactive tool for joint use by spina bifida patients and their urologists to identify patients interested in addressing their urinary and fecal incontinence and establish continence goal(s) they would like to achieve. To date, no such tool exists for use by spina bifida patients or urologists. This represents a major paradigm shift in the urologic care of pediatric SB patients. It will give children and families a voice in setting their personal goals for urinary and fecal incontinence, rather than relying on physicians' traditional clinical targets (e.g., absence of urinary incontinence, 4-hour dry interval). These traditional views fail to reflect the full patient experience of their ailment by underestimating symptoms and prioritizing only the most severe. This study represents the first time that such a process will be formalized before initiating urological therapy in children with SB (Aim 2). Additionally, this tool may help rule out interventions with a low chance of achieving desired goals and allow for a recalibration of unrealistic goals. The app will be useful for any child, regardless of urinary and fecal incontinence treatment history or underlying bladder pathology, as it will help describe personalized clinical treatment goals based on urinary incontinence, a characteristic all these patients share. This study will also capture the health-related quality of life (HRQOL) impact of urinary and fecal incontinence improvement regardless of the treatment, whether behavioral, medical or surgical, many of which are available to patients regardless of age. A systematic therapeutic goal-setting tool will help in bringing precision medicine to the SB population.

DETAILED DESCRIPTION:
Phase 1: Stakeholder Group. The investigators will engage 30 dyads of children and adolescents with spina bifida aged 8-17 years old, who experienced any urinary and fecal incontinence in the past 4 weeks, and their caregivers in the exploration phase. These children and adolescents will be identified from among spina bifida patients receiving care from pediatric urology providers at Riley Hospital for Children, Indiana University Health. As part of the exploration process, it is important to include patients that reflect the varied life experiences of those impacted by spina bifida. Therefore, the investigators will aim to include children and adolescents with a range of physical and cognitive developmental delays. Groups will be separated by gender to facilitate discussion and elicit any gender-specific urinary incontinence goals. The patient engagement core will create a smartphone-based "Day in the Life" diary toolkit that will be provided to the stakeholder group. The stakeholders will be asked to self-report their experiences and perspectives as they relate to being a child or adolescent with spina bifida and urinary and fecal incontinence, or taking care of someone with spina bifida with urinary incontinence. Stakeholders will be asked to respond using video to various prompts such as documenting a typical day in their life, sharing their experiences. After completing the requested tasks, stakeholders will return the toolkit to the patient engagement. These self-reporting tools will be designed to be as usable as possible by as many participants as possible, taking into account common barriers caused by this condition, and relying on caregivers, as needed, to administer the tools. Investigators anticipate that the kit will take approximately 3 hours to complete. Through analysis and translation of the diaries and video, the patient engagement core will identify insights into patient-centered UI goals and areas of opportunity for design solutions. These identified opportunity spaces will inform the work for Phase Two, the creation phase.

Phase 2: In order to achieve a holistic and sustainable intervention, it is crucial that the investigators work with an interdisciplinary team that include designers, researchers, patients, family members, other caregivers, and health care providers in the process of creating the intervention. Therefore, the investigators will invite 8-10 of the dyads from Phase One to participate as members of the Co-Design Panel which will be brought together to participate in a 2-4 hour co-design session. During this session, designers will share the insights gained from Phase One work. Panel participants will be asked to help refine these insights to define domains of patient-centered urinary incontinence goals. From there, the Co-Design Panel will work to generate solutions for a tool to facilitate goal-setting and follow-up related to these domains (i.e., the tool, or app). This will be done through a series of generative, prototyping exercises with participants. For example, the group could work in small teams to generate ideas for their ideal goal-setting tool and then use sketches, storyboards, building materials like foam core, or verbal story-telling to prototype these ideas. The options for prototyping will be diverse to accommodate a spectrum of physical and cognitive abilities. These prototypes can then be used to generate discussion among the Co-Design Panel, which will further refine the ideal aspects of the app from the perspective of children and adolescents with SB and their caregivers.

The Physician Panel will then be invited to respond to a prototype of the app and give their input on how it can be improved to best fit into clinic workflow, address physician preferences, and work for a variety of patient-physician scenarios. These responses will be gathered through structured in-person interviews.

Phase 3: The investigators will ask patient/caregiver dyads with spina bifida (N=8), who were not part of the Co-Design Panel in Phase Two, to utilize the tool in conjunction with their pediatric urologist during a pediatric urology clinic visit at Riley Hospital. The investigators will comply with all IRB requirements at the study institution for the inclusion of patients in research, including obtaining the necessary consents/assents.

Testing Process. Following the clinic visit, the patient/caregiver will participate in Cognitive Interviews. They will be asked to describe their impressions of the prototype app through the use of scripted verbal probes ("What do you think is being represented here?" "Describe what you would do next.") and spontaneous probes ("What about this picture/sentence/etc., makes you feel that way?"), the investigators will determine if the prototype app is functioning as expected, or any key elements were missed. The investigators will also ask for feedback from the urologists on how well the tool functioned within the clinic setting to help in this iterative validation process. This will be accomplished by conducting interviews with approximately 6 physicians.

Phase 4: The investigators will recruit children and adolescents with SB (8-17 years old) who are followed at Riley Hospital Pediatric Urology Outpatient Clinic and their primary caregiver. The primary caregiver must be the patient's legal guardian. Well over 200 children and adolescents with SB are seen at this facility annually. Each week, a research assistant (RA) will be given a list of SB patients within the desired age range who have an upcoming appointment in two settings: the Pediatric Urology Clinic or the multidisciplinary Spina Bifida clinic. The RA will approach the patient and their primary caregiver upon arrival at the clinic appointment to gauge their interest in study participation. If the dyad indicates potential interest, the RA will take them to a private area to further discuss the details of the study, determine eligibility, and then obtain consent from the legal caregiver and assent from the patient wishing to enroll in the study. Over a 12-month period, the investigators will enroll 92 children and adolescents with SB and their primary caregivers. After enrollment in the study, the RA will administer the app, and collect baseline data regarding self-reported urinary and fecal incontinence and HRQOL. The patient and their caregiver will then meet with their urologist for the scheduled clinic appointment. After being enrolled at baseline, participants will continue with standard care for 12 months (while completing UI, HRQOL, and other questionnaires), at which point the app is introduced and the goal is set, and then they are followed for another 12 months. The urologist will be provided with the completed app and will utilize this tool to verify/discuss the goal selected, and then discuss plans for treatment in order to achieve this goal. Goal attainment, UI, and HRQOL will be assessed at 6 and 12 months after the app is introduced. Children with SB are typically seen in the outpatient clinic every 6-12 months. Therefore, these follow-up assessments will occur in-person at a clinic appointment, or, if not possible, investigators will contact the participant by telephone to notify them that an email link to a secure website to complete the necessary assessments will be sent. To minimize loss to follow-up, investigators will ask for 3 different phone numbers with at least one being a landline (if available). Investigators will also ask for two email addresses. Up to 3 attempts will be made to reach participants.

ELIGIBILITY:
Inclusion Criteria:

* Spina bifida
* 8-17 years old
* Followed at Riley Hospital Pediatric Urology Outpatient Clinic
* Primary caregiver is patient's legal guardian
* Urinary incontinence in the past 4 weeks
* Fecal incontinence in the past 4 weeks
* Normal to mildly impaired cognitive development
* English language literacy
* Intent to receive care at the Riley Pediatric Urology Clinic for th extent of the study

The physician panel will be composed of pediatric urologists.

Exclusion Criteria:

* Children with significant cognitive impairment, as they will not be able to express their urinary and fecal incontinence goals.
* Patients who underwent a genitourinary procedure or a bowel procedure in the past 4 weeks, since these patients are often temporarily catheterized and therefore not experiencing their typical level of urinary and fecal incontinence.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
SB-specific HRQOL | 2 years
  The primary outcome, SB-specific HRQOL, will be evaluated using the validated 10-item QUAlity of Life ASsessment in Children/Teenagers (QUALAS-C/T) questionnaire. Scores range from 0 to 100, with higher scores signifying better HRQOL.

SECONDARY OUTCOMES:
Shared decision making | 2 years
  SDM will be evaluated with the 9-item Shared Decision Making questionnaire (SDM-Q-9). Scores range from 0 to 100, with higher scores signifying better SDM.
Patient-provider communication | 2 years
  This will be evaluated with a 13-item Health Care Climate Questionnaire (HCCQ). Scores range from 1 to 7, with higher scores signifying better patient-provider communication.
UI Goal selection and attainement | 2 years
  Goals and goal attainment will be assessed using the MyGoal tool. Patients who select a UI goal will be considered to be concerned about UI and offered UI treatments. Those who do not select a UI goal will be considered not to be concerned. Self-reported goal attainment will be categorized as: attained, not attained, and goal initially not identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liptak GS, Garver K, Dosa NP. Spina bifida grown up. J Dev Behav Pediatr. 2013 Apr;34(3):206-15. doi: 10.1097/DBP.0b013e31828c5f88. PMID 23572172
- [Background] Woodhouse CR, Neild GH, Yu RN, Bauer S. Adult care of children from pediatric urology. J Urol. 2012 Apr;187(4):1164-71. doi: 10.1016/j.juro.2011.12.011. Epub 2012 Feb 14. PMID 22335866
- [Background] Stohrer M, Blok B, Castro-Diaz D, Chartier-Kastler E, Del Popolo G, Kramer G, Pannek J, Radziszewski P, Wyndaele JJ. EAU guidelines on neurogenic lower urinary tract dysfunction. Eur Urol. 2009 Jul;56(1):81-8. doi: 10.1016/j.eururo.2009.04.028. Epub 2009 Apr 21. PMID 19403235
- [Background] Malone PS, Wheeler RA, Williams JE. Continence in patients with spina bifida: long term results. Arch Dis Child. 1994 Feb;70(2):107-10. doi: 10.1136/adc.70.2.107. PMID 8129429
- [Background] Whittam B, Szymanski K, Misseri R, Carroll A, Kaefer M, Rink R, Cain M. Long-term fate of the bladder after isolated bladder neck procedure. J Pediatr Urol. 2014 Oct;10(5):886-91. doi: 10.1016/j.jpurol.2013.12.022. Epub 2014 Jan 25. PMID 24517903
- [Background] Herndon CD, Rink RC, Shaw MB, Simmons GR, Cain MP, Kaefer M, Casale AJ. The Indiana experience with artificial urinary sphincters in children and young adults. J Urol. 2003 Feb;169(2):650-4; discussion 654. doi: 10.1097/01.ju.0000047320.28201.9d. PMID 12544336
- [Background] Tapia CI, Khalaf K, Berenson K, Globe D, Chancellor M, Carr LK. Health-related quality of life and economic impact of urinary incontinence due to detrusor overactivity associated with a neurologic condition: a systematic review. Health Qual Life Outcomes. 2013 Jan 31;11:13. doi: 10.1186/1477-7525-11-13. PMID 23369111
- [Background] Lemelle JL, Guillemin F, Aubert D, Guys JM, Lottmann H, Lortat-Jacob S, Mouriquand P, Ruffion A, Moscovici J, Schmitt M. Quality of life and continence in patients with spina bifida. Qual Life Res. 2006 Nov;15(9):1481-92. doi: 10.1007/s11136-006-0032-x. Epub 2006 Oct 11. PMID 17033913
- [Background] Vu Minh Arnell M, Seljee Svedberg K, Lindehall B, Moller A, Abrahamsson K. Health-related quality of life compared to life situation and incontinence in adults with myelomeningocele: is SF-36 a reliable tool? J Pediatr Urol. 2013 Oct;9(5):559-66. doi: 10.1016/j.jpurol.2013.05.005. Epub 2013 Jun 12. PMID 23769200
- [Background] Olesen JD, Kiddoo DA, Metcalfe PD. The association between urinary continence and quality of life in paediatric patients with spina bifida and tethered cord. Paediatr Child Health. 2013 Aug;18(7):e32-8. PMID 24421717
- [Background] MacNeily AE, Jafari S, Scott H, Dalgetty A, Afshar K. Health related quality of life in patients with spina bifida: a prospective assessment before and after lower urinary tract reconstruction. J Urol. 2009 Oct;182(4 Suppl):1984-91. doi: 10.1016/j.juro.2009.02.060. Epub 2009 Aug 20. PMID 19695599
- [Background] Ramachandra P, Palazzi KL, Skalsky AJ, Marietti S, Chiang G. Shunted hydrocephalus has a significant impact on quality of life in children with spina bifida. PM R. 2013 Oct;5(10):825-31. doi: 10.1016/j.pmrj.2013.05.011. Epub 2013 May 22. PMID 23707568
- [Background] Waters E, Davis E, Ronen GM, Rosenbaum P, Livingston M, Saigal S. Quality of life instruments for children and adolescents with neurodisabilities: how to choose the appropriate instrument. Dev Med Child Neurol. 2009 Aug;51(8):660-9. doi: 10.1111/j.1469-8749.2009.03324.x. PMID 19627340
- [Background] Szymanski KM, Wheeler DC, Mucci LA. Fish consumption and prostate cancer risk: a review and meta-analysis. Am J Clin Nutr. 2010 Nov;92(5):1223-33. doi: 10.3945/ajcn.2010.29530. Epub 2010 Sep 15. PMID 20844069
- [Background] Szymanski KM, Oliveira LM, Silva A, Retik AB, Nguyen HT. Analysis of indications for ureteral reimplantation in 3738 children with vesicoureteral reflux: a single institutional cohort. J Pediatr Urol. 2011 Dec;7(6):601-10. doi: 10.1016/j.jpurol.2011.06.002. Epub 2011 Jul 7. PMID 21741318
- [Background] Szymanski KM, Wei JT, Dunn RL, Sanda MG. Development and validation of an abbreviated version of the expanded prostate cancer index composite instrument for measuring health-related quality of life among prostate cancer survivors. Urology. 2010 Nov;76(5):1245-50. doi: 10.1016/j.urology.2010.01.027. Epub 2010 Mar 28. PMID 20350762
- [Background] Chang P, Szymanski KM, Dunn RL, Chipman JJ, Litwin MS, Nguyen PL, Sweeney CJ, Cook R, Wagner AA, DeWolf WC, Bubley GJ, Funches R, Aronovitz JA, Wei JT, Sanda MG. Expanded prostate cancer index composite for clinical practice: development and validation of a practical health related quality of life instrument for use in the routine clinical care of patients with prostate cancer. J Urol. 2011 Sep;186(3):865-72. doi: 10.1016/j.juro.2011.04.085. Epub 2011 Jul 23. PMID 21788038
- [Background] Szymanski KM, Bitzan M, Capolicchio JP. Is retroperitoneoscopy the gold standard for endoscopic nephrectomy in children on peritoneal dialysis? J Urol. 2010 Oct;184(4 Suppl):1631-7. doi: 10.1016/j.juro.2010.04.019. Epub 2010 Aug 21. PMID 20728139
- [Background] Szymanski KM, Al-Said AN, Pippi Salle JL, Capolicchio JP. Do infants with mild prenatal hydronephrosis benefit from screening for vesicoureteral reflux? J Urol. 2012 Aug;188(2):576-81. doi: 10.1016/j.juro.2012.04.017. Epub 2012 Jun 15. PMID 22704090
- [Background] Szymanski KM, St-Cyr D, Alam T, Kassouf W. External stoma and peristomal complications following radical cystectomy and ileal conduit diversion: a systematic review. Ostomy Wound Manage. 2010 Jan 1;56(1):28-35. PMID 20093715
- [Background] Wheeler DC, Szymanski KM, Black A, Nelson DE. Applying strategies from libertarian paternalism to decision making for prostate specific antigen (PSA) screening. BMC Cancer. 2011 Apr 21;11:148. doi: 10.1186/1471-2407-11-148. PMID 21510865
- [Background] Azhar RA, Szymanski KM, Lemercier E, Valenti D, Andonian S, Anidjar M. Visceral organ-to-percutaneous tract distance is shorter when patients are placed in the prone position on bolsters compared with the supine position. J Endourol. 2011 Apr;25(4):687-90. doi: 10.1089/end.2010.0547. Epub 2011 Mar 25. PMID 21438689
- [Background] Ghane Sharbaf F, Bitzan M, Szymanski KM, Bell LE, Gupta I, Tchervenkov J, Capolicchio JP. Native nephrectomy prior to pediatric kidney transplantation: biological and clinical aspects. Pediatr Nephrol. 2012 Jul;27(7):1179-88. doi: 10.1007/s00467-012-2115-y. Epub 2012 Feb 26. PMID 22366876
- [Background] Mansure JJ, Nassim R, Chevalier S, Szymanski K, Rocha J, Aldousari S, Kassouf W. A novel mechanism of PPAR gamma induction via EGFR signalling constitutes rational for combination therapy in bladder cancer. PLoS One. 2013;8(2):e55997. doi: 10.1371/journal.pone.0055997. Epub 2013 Feb 8. PMID 23409107
- [Background] Violette P, Abourbih S, Szymanski KM, Tanguay S, Aprikian A, Matthews K, Brimo F, Kassouf W. Solitary solid renal mass: can we predict malignancy? BJU Int. 2012 Dec;110(11 Pt B):E548-52. doi: 10.1111/j.1464-410X.2012.11245.x. Epub 2012 May 22. PMID 22612453
- [Background] Violette PD, Szymanski KM, Anidjar M, Andonian S. Factors determining fluoroscopy time during ureteroscopy. J Endourol. 2011 Dec;25(12):1837-40. doi: 10.1089/end.2011.0204. Epub 2011 Sep 9. PMID 21905847
- [Background] Szymanski KM, Misseri R, Whittam B, Raposo SM, King SJ, Kaefer M, Rink RC, Cain MP. QUAlity of Life Assessment in Spina bifida for Adults (QUALAS-A): development and international validation of a novel health-related quality of life instrument. Qual Life Res. 2015 Oct;24(10):2355-64. doi: 10.1007/s11136-015-0988-5. Epub 2015 Apr 12. PMID 25863685
- [Background] Szymanski KM, Misseri R, Whittam B, Yang DY, Raposo SM, King SJ, Kaefer M, Rink RC, Cain MP. Quality of Life Assessment in Spina Bifida for Children (QUALAS-C): Development and Validation of a Novel Health-related Quality of Life Instrument. Urology. 2016 Jan;87:178-84. doi: 10.1016/j.urology.2015.09.027. Epub 2015 Oct 9. PMID 26456744
- [Background] Szymanski KM, Misseri R, Whittam B, Adams CM, Kirkegaard J, King S, Kaefer M, Rink RC, Cain MP. Mortality after bladder augmentation in children with spina bifida. J Urol. 2015 Feb;193(2):643-8. doi: 10.1016/j.juro.2014.07.101. Epub 2014 Jul 27. PMID 25072178
- [Background] Szymanski KM, Misseri R, Whittam B, Amstutz S, Kaefer M, Rink RC, Cain MP. Cutting for stone in augmented bladders-what is the risk of recurrence and is it impacted by treatment modality? J Urol. 2014 May;191(5):1375-80. doi: 10.1016/j.juro.2013.11.057. Epub 2013 Dec 5. PMID 24316089
- [Background] Szymanski KM, Keenan A, Cain MP, Waseem S, Kaefer M. A novel colonoscopic approach for the management of a Malone antegrade continence enema channel, which cannot be catheterized in the immediate postoperative period: a case report. Urology. 2014 Dec;84(6):1490-1. doi: 10.1016/j.urology.2014.07.047. Epub 2014 Oct 11. PMID 25306482
- [Background] Calaway AC, Whittam B, Szymanski KM, Misseri R, Kaefer M, Rink RC, Karymazn B, Cain MP. Multicystic dysplastic kidney: is an initial voiding cystourethrogram necessary? Can J Urol. 2014 Oct;21(5):7510-4. PMID 25347379
- [Background] Whittam BM, Calaway A, Szymanski KM, Carroll AE, Misseri R, Kaefer M, Rink RC, Karmazyn B, Cain MP. Ultrasound diagnosis of multicystic dysplastic kidney: is a confirmatory nuclear medicine scan necessary? J Pediatr Urol. 2014 Dec;10(6):1059-62. doi: 10.1016/j.jpurol.2014.03.011. Epub 2014 May 2. PMID 24909606
- [Background] Szymanski KM, Tabib CH, Idrees MT, Cain MP. Synchronous perivesical and renal malignant rhabdoid tumor in a 9-year-old boy: a case report and review of literature. Urology. 2013 Nov;82(5):1158-60. doi: 10.1016/j.urology.2013.04.050. Epub 2013 Jul 3. PMID 23830079
- [Background] Chan KH, Szymanski KM, Li X, Ofner S, Flack C, Judge B, Whittam B, Misseri R, Kaefer M, Rink RC, Cain MP. Effect of baseline obesity and postoperative weight gain on the risk of channel revision following continent catheterizable urinary channel surgery. J Pediatr Urol. 2016 Aug;12(4):249.e1-7. doi: 10.1016/j.jpurol.2016.05.021. Epub 2016 Jun 11. PMID 27480466
- [Background] Whittam BM, Szymanski KM, Flack C, Misseri R, Kaefer M, Rink RC, Cain MP. A comparison of the Monti and spiral Monti procedures: A long-term analysis. J Pediatr Urol. 2015 Jun;11(3):134.e1-6. doi: 10.1016/j.jpurol.2014.12.013. Epub 2015 Mar 25. PMID 25936690
- [Background] Szymanski KM, Whittam B, Misseri R, Flack CK, Hubert KC, Kaefer M, Rink RC, Cain MP. Long-term outcomes of catheterizable continent urinary channels: What do you use, where you put it, and does it matter? J Pediatr Urol. 2015 Aug;11(4):210.e1-7. doi: 10.1016/j.jpurol.2015.05.002. Epub 2015 May 30. PMID 26071074
- [Background] Casey JT, Zhang M, Chan KH, Szymanski KM, Judge B, Whittam B, Kaefer M, Misseri R, Rink RC, Cain MP. Does endoscopy of difficult to catheterize channels spare some patients from formal open revision? J Pediatr Urol. 2016 Aug;12(4):248.e1-6. doi: 10.1016/j.jpurol.2016.04.030. Epub 2016 May 26. PMID 27270068
- [Background] Szymanski KM, Whittam B, Misseri R, Chan KH, Flack CK, Kaefer M, Rink RC, Cain MP. A case of base rate bias, or are adolescents at a higher risk of developing complications after catheterizable urinary channel surgery? J Pediatr Urol. 2017 Apr;13(2):184.e1-184.e6. doi: 10.1016/j.jpurol.2016.12.002. Epub 2017 Jan 11. PMID 28159526
- [Background] Large T, Szymanski KM, Whittam B, Misseri R, Chan KH, Kaefer M, Rink RC, Cain MP. Ambulatory patients with spina bifida are 50% more likely to be fecally continent than non-ambulatory patients, particularly after a MACE procedure. J Pediatr Urol. 2017 Feb;13(1):60.e1-60.e6. doi: 10.1016/j.jpurol.2016.06.019. Epub 2016 Aug 24. PMID 27614699
- [Background] Szymanski KM, Misseri R, Whittam B, Lingeman JE, Amstutz S, Ring JD, Kaefer M, Rink RC, Cain MP. Bladder stones after bladder augmentation are not what they seem. J Pediatr Urol. 2016 Apr;12(2):98.e1-6. doi: 10.1016/j.jpurol.2015.06.021. Epub 2015 Sep 25. PMID 26455637
- [Background] Hubert KC, Large T, Leiser J, Judge B, Szymanski K, Whittam B, Kaefer M, Misseri R, Rink R, Cain MP. Long-term renal functional outcomes after primary gastrocystoplasty. J Urol. 2015 Jun;193(6):2079-84. doi: 10.1016/j.juro.2014.12.088. Epub 2015 Jan 3. PMID 25562446
- [Background] Szymanski KM, Rink RC, Whittam B, Ring JD, Misseri R, Kaefer M, Cain MP. Long-term outcomes of the Kropp and Salle urethral lengthening bladder neck reconstruction procedures. J Pediatr Urol. 2016 Dec;12(6):403.e1-403.e7. doi: 10.1016/j.jpurol.2016.06.011. Epub 2016 Jul 26. PMID 27687531
- [Background] Szymanski KM, Cain MP, Hardacker TJ, Misseri R. How successful is the transition to adult urology care in spina bifida? A single center 7-year experience. J Pediatr Urol. 2017 Feb;13(1):40.e1-40.e6. doi: 10.1016/j.jpurol.2016.09.020. Epub 2016 Nov 9. PMID 27979598
- [Background] Roth JD, Misseri R, Cain MP, Szymanski KM. Mobility, hydrocephalus and quality of erections in men with spina bifida. J Pediatr Urol. 2017 Jun;13(3):264.e1-264.e6. doi: 10.1016/j.jpurol.2016.12.004. Epub 2017 Jan 11. PMID 28111207
- [Background] Szymanski KM, Misseri R, Whittam B, Large T, Cain MP. Current opinions regarding care of the mature pediatric urology patient. J Pediatr Urol. 2015 Oct;11(5):251.e1-4. doi: 10.1016/j.jpurol.2015.05.020. Epub 2015 Jun 21. PMID 26148437
- [Background] Strine AC, Misseri R, Szymanski KM, Kaefer M, Rhee AC, Hillier K, Rink RC, Cain MP. Assessing health related benefit after reconstruction for urinary and fecal incontinence in children: a parental perspective. J Urol. 2015 Jun;193(6):2073-8. doi: 10.1016/j.juro.2014.12.089. Epub 2015 Jan 3. PMID 25562445
- [Background] Szymanski KM, Misseri R, Whittam B, Kaefer M, Rink RC, Cain MP. Quantity, Not Frequency, Predicts Bother with Urinary Incontinence and its Impact on Quality of Life in Adults with Spina Bifida. J Urol. 2016 Apr;195(4 Pt 2):1263-9. doi: 10.1016/j.juro.2015.07.108. Epub 2016 Feb 28. PMID 26926556
- [Background] Szymanski KM, Cain MP, Whittam B, Kaefer M, Rink RC, Misseri R. All Incontinence is Not Created Equal: Impact of Urinary and Fecal Incontinence on Quality of Life in Adults with Spina Bifida. J Urol. 2017 Mar;197(3 Pt 2):885-891. doi: 10.1016/j.juro.2016.08.117. Epub 2017 Jan 26. PMID 28131501
- [Background] Snow-Lisy DC, Yerkes EB, Cheng EY. Update on Urological Management of Spina Bifida from Prenatal Diagnosis to Adulthood. J Urol. 2015 Aug;194(2):288-96. doi: 10.1016/j.juro.2015.03.107. Epub 2015 Apr 1. PMID 25839383
- [Background] Metcalfe PD, Cain MP, Kaefer M, Gilley DA, Meldrum KK, Misseri R, King SJ, Casale AJ, Rink RC. What is the need for additional bladder surgery after bladder augmentation in childhood? J Urol. 2006 Oct;176(4 Pt 2):1801-5; discussion 1805. doi: 10.1016/j.juro.2006.03.126. PMID 16945653
- [Background] Salle JL, McLorie GA, Bagli DJ, Khoury AE. Urethral lengthening with anterior bladder wall flap (Pippi Salle procedure): modifications and extended indications of the technique. J Urol. 1997 Aug;158(2):585-90. doi: 10.1097/00005392-199708000-00092. PMID 9224369
- [Background] Murray CB, Holmbeck GN, Ros AM, Flores DM, Mir SA, Varni JW. A longitudinal examination of health-related quality of life in children and adolescents with spina bifida. J Pediatr Psychol. 2015 May;40(4):419-30. doi: 10.1093/jpepsy/jsu098. Epub 2014 Nov 29. PMID 25434043
- [Background] Sawin KJ, Bellin MH. Quality of life in individuals with spina bifida: a research update. Dev Disabil Res Rev. 2010;16(1):47-59. doi: 10.1002/ddrr.96. PMID 20419771
- [Background] Lloyd JC, Nseyo U, Madden-Fuentes RJ, Ross SS, Wiener JS, Routh JC. Reviewing definitions of urinary continence in the contemporary spina bifida literature: a call for clarity. J Pediatr Urol. 2013 Oct;9(5):567-74. doi: 10.1016/j.jpurol.2013.02.006. Epub 2013 Mar 16. PMID 23507290
- [Background] Kiresuk TJ, Sherman RE. Goal attainment scaling: A general method for evaluating comprehensive community mental health programs. Community Ment Health J. 1968 Dec;4(6):443-53. doi: 10.1007/BF01530764. PMID 24185570
- [Background] Hullfish KL, Bovbjerg VE, Gurka MJ, Steers WD. Surgical versus nonsurgical treatment of women with pelvic floor dysfunction: patient centered goals at 1 year. J Urol. 2008 Jun;179(6):2280-5; discussion 2285. doi: 10.1016/j.juro.2008.01.147. Epub 2008 Apr 18. PMID 18423762
- [Background] Anderson CB, Rapkin B, Reaves BC, Sun AJ, Morganstern B, Dalbagni G, Donat M, Herr HW, Laudone VP, Bochner BH. Idiographic quality of life assessment before radical cystectomy. Psychooncology. 2017 Feb;26(2):206-213. doi: 10.1002/pon.4025. Epub 2015 Nov 30. PMID 26620583
- [Background] Vroland-Nordstrand K, Eliasson AC, Jacobsson H, Johansson U, Krumlinde-Sundholm L. Can children identify and achieve goals for intervention? A randomized trial comparing two goal-setting approaches. Dev Med Child Neurol. 2016 Jun;58(6):589-96. doi: 10.1111/dmcn.12925. Epub 2015 Sep 16. PMID 26374194
- [Background] Missiuna C, DeMatteo C, Hanna S, Mandich A, Law M, Mahoney W, Scott L. Exploring the use of cognitive intervention for children with acquired brain injury. Phys Occup Ther Pediatr. 2010 Aug;30(3):205-19. doi: 10.3109/01942631003761554. PMID 20608858
- [Background] Speth L, Janssen-Potten Y, Rameckers E, Defesche A, Winkens B, Becher J, Smeets R, Vles H. Effects of botulinum toxin A and/or bimanual task-oriented therapy on upper extremity activities in unilateral Cerebral Palsy: a clinical trial. BMC Neurol. 2015 Aug 19;15:143. doi: 10.1186/s12883-015-0404-3. PMID 26286662
- [Background] Constand MK, MacDermid JC. Applications of the International Classification of Functioning, Disability and Health in goal-setting practices in healthcare. Disabil Rehabil. 2014;36(15):1305-14. doi: 10.3109/09638288.2013.845256. Epub 2013 Oct 23. PMID 24151819
- [Background] Pasch L, He SY, Huddleston H, Cedars MI, Beshay A, Zane LT, Shinkai K. Clinician vs Self-ratings of Hirsutism in Patients With Polycystic Ovarian Syndrome: Associations With Quality of Life and Depression. JAMA Dermatol. 2016 Jul 1;152(7):783-8. doi: 10.1001/jamadermatol.2016.0358. PMID 26942548
- [Background] Hinami K, Alkhalil A, Chouksey S, Chua J, Trick WE. Clinical significance of physical symptom severity in standardized assessments of patient reported outcomes. Qual Life Res. 2016 Sep;25(9):2239-43. doi: 10.1007/s11136-016-1261-2. Epub 2016 Mar 15. PMID 26980417
- [Background] Collins FS, Varmus H. A new initiative on precision medicine. N Engl J Med. 2015 Feb 26;372(9):793-5. doi: 10.1056/NEJMp1500523. Epub 2015 Jan 30. PMID 25635347
- [Background] Matheson GO, Pacione C, Shultz RK, Klugl M. Leveraging human-centered design in chronic disease prevention. Am J Prev Med. 2015 Apr;48(4):472-9. doi: 10.1016/j.amepre.2014.10.014. Epub 2015 Feb 18. PMID 25700655
- [Background] Searl MM, Borgi L, Chemali Z. It is time to talk about people: a human-centered healthcare system. Health Res Policy Syst. 2010 Nov 26;8:35. doi: 10.1186/1478-4505-8-35. PMID 21110859
- [Background] Domecq JP, Prutsky G, Elraiyah T, Wang Z, Nabhan M, Shippee N, Brito JP, Boehmer K, Hasan R, Firwana B, Erwin P, Eton D, Sloan J, Montori V, Asi N, Dabrh AM, Murad MH. Patient engagement in research: a systematic review. BMC Health Serv Res. 2014 Feb 26;14:89. doi: 10.1186/1472-6963-14-89. PMID 24568690
- [Background] Ravens-Sieberer U, Auquier P, Erhart M, Gosch A, Rajmil L, Bruil J, Power M, Duer W, Cloetta B, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. The KIDSCREEN-27 quality of life measure for children and adolescents: psychometric results from a cross-cultural survey in 13 European countries. Qual Life Res. 2007 Oct;16(8):1347-56. doi: 10.1007/s11136-007-9240-2. Epub 2007 Aug 1. PMID 17668292
- [Background] Muthen B, Shedden K. Finite mixture modeling with mixture outcomes using the EM algorithm. Biometrics. 1999 Jun;55(2):463-9. doi: 10.1111/j.0006-341x.1999.00463.x. PMID 11318201
- [Background] Proust C, Jacqmin-Gadda H. Estimation of linear mixed models with a mixture of distribution for the random effects. Comput Methods Programs Biomed. 2005 May;78(2):165-73. doi: 10.1016/j.cmpb.2004.12.004. PMID 15848271
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Zappitelli M, Parvex P, Joseph L, Paradis G, Grey V, Lau S, Bell L. Derivation and validation of cystatin C-based prediction equations for GFR in children. Am J Kidney Dis. 2006 Aug;48(2):221-30. doi: 10.1053/j.ajkd.2006.04.085. PMID 16860187
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Boulet SL, Yang Q, Mai C, Kirby RS, Collins JS, Robbins JM, Meyer R, Canfield MA, Mulinare J; National Birth Defects Prevention Network. Trends in the postfortification prevalence of spina bifida and anencephaly in the United States. Birth Defects Res A Clin Mol Teratol. 2008 Jul;82(7):527-32. doi: 10.1002/bdra.20468. PMID 18481813
- [Background] Elkoshy M, Szymanski KM, Morehouse D, Anidjar M, Andonian S. Shock-wave lithotripsy retreatment rates among three different lithotripters. UroToday Int. June 2012 2012;5(3):18.
- [Background] Giacomin J. What Is Human Centred Design? The Design Journal. 2014/12/01 2014;17(4):606-623.
- [Background] Sanematsu H, Wiehe S. Learning to look: Design in health services research. Touchpoint. 2014;July:TP06-02P82.
- [Background] Jones JHC, Thornley DG. Conference on Design Methods. Oxford, New York,: Pergamon Press; 1963.
- [Background] Sanematsu H, Wiehe S. How do you do? Design research methods and the
- [Background] Sanematsu H. 53. Fun with Facebook: The Impact of Focus Groups on the Development of Awareness Campaigns for Adolescent Health. Journal of Adolescent Health. January 2011 2011;48(2):S44-S45.
- [Background] Nielsen J. Estimating the number of subjects needed for a thinking aloud test. Int J Human-Computer Studies. 1994;41:385-397.
- [Background] Stickdorn M, Schneider J. This is Service Design Thinking. Basics - Tools - Cases. Amsterdam: BIS Publishers; 2011.
- [Background] Singer JD, Willett JB. Applied longitudinal data analysis : modeling change and event occurrence. Oxford ; New York: Oxford University Press; 2003.
- See also: Hasso Plattner Institute of Design. bootcamp bootleg Accessed March 24, 2015. — https://dschool.stanford.edu/resources/the-bootcamp-bootleg